





## UNIVERSITETI I MJEKËSISË, TIRANË KËSHILLI I ETIKËS

Nr. 3232 prot.

Tiránë, më <u>06.12</u>.2024

Lënda:

Njoftim mbi miratimin e Studimit/Projektit kërkimor

## MARTIOLA KOLA FAKULTETI I MJEKËSISË UNIVERSITETI I MJEKËSISË, TIRANË

Kětu

E nderuar,

Pasi kemi marrë në shqyrtim aplikimin tuaj "NLR, si një parashikues i rëndësishëm në pacientët Post ACS", ju njoftojmë se projekti juaj kërkimor është miratuar nga Këshilli i Etikës pranë Universitetit të Mjekësisë Tiranë.

Duke ju falënderuar për bashkëpunimin,

